CLINICAL TRIAL: NCT03964584
Title: Evaluation of the Neurological and Psychiatric Adverse Events of Dolutegravir and Bictegravir in Real Life (NEPALE)
Brief Title: Evaluation of the Neurological and Psychiatric Adverse Events of Dolutegravir and Bictegravir in Real Life
Acronym: NEPALE
Status: Withdrawn | Type: Observational
Why Stopped: Low scientific relevance due to the marketing of new treatments, and expected inclusion difficulties
Sponsor: Fondation Ophtalmologique Adolphe de Rothschild (Network)
Responsible Party: Sponsor
Other Study IDs: AMR_2019_1
Record Dates: First submitted 2019-05-24; First posted 2019-05-28 (Actual); Last update posted 2020-02-27 (Actual); Status verified 2020-02

CONDITIONS: HIV+ Patients
Keywords: dolutegravir; dictegravir; Neurological disorder; Psychiatric disorder; HIV integrase Inhibitors; Adverse drug event
MeSH Terms: conditions — Nervous System Diseases; Mental Disorders; Drug-Related Side Effects and Adverse Reactions

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: assessment of neurological and psychiatric disorders by self-administered questionnaires — Patients will be included on the day dolutegravir or bictegravir is prescribed. Neurological and psychiatric disorders will be assessed using self-administered questionnaires, at inclusion, one month, three months and six months.

SUMMARY:
The neurological and psychiatric adverse effects of antiretroviral drugs is a concern for clinicians and people living with HIV. In addition, clinical trials conducted prior to market authorization often have stric inclusion and exclusion criteria in terms of age, co-morbidity or co-medication, and the patients included in the studies are not always representative of the population for whom the drugs will be prescribed in real life. We propose a prospective cohort study to assess the occurrence of neurological and psychiatric adverse events in HIV+ patients starting an association with dolutegravir or bictegravir.

Patients will be included on the day dolutegravir or bictegravir is prescribed. Neurological and psychiatric disorders will be assessed using self-administered questionnaires, at inclusion, one month, three months and six months.

ELIGIBILITY:
Inclusion criteria:

* Age ≥ 18 years
* HIV-infected
* Initiation or modification of antiretroviral therapy, and starting a therapeutic combination including dolutegravir or bictegravir

Exclusion criteria:

* Intolerance to dolutegravir or bictegravir
* Addiction to a psychoactive product (drugs or medications) with the exception of amyl nitriles ("poppers") and occasional recreational cannabis
* Alcohol consumption >10 standard drinks/week
* Active HCV coinfection
* Pregnant or breastfeeding woman

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: HIV infected patients who need to initiate or modify antiretroviral therapy, and starting a combination of antiretroviral agents including dolutegravir or bictegravir.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2019-09-01 (Actual); Primary Completion 2019-09-01 (Actual); Study Completion 2019-09-01 (Actual)

PRIMARY OUTCOMES:
The presence of at least one of the following neurological or psychiatric disorders | 6 months
  * depression, defined by a CES-D score ≥ 17 for men and ≥ 23 for women
  * anxiety, defined by a STAI score ≥ 56 (high anxiety); a score > 65 indicating very high anxiety;
  * pathological fatigue, defined by a score on the EMIF-SEP scale ≥ 45/100;
  * presence of a neurological symptom identified by the QES questionnaire.

IPD SHARING:
Plan to Share IPD: No